CLINICAL TRIAL: NCT02223351
Title: A Single-centre, Open-label, Randomised, Crossover, Drug-drug Interaction Study to Investigate the Effect of a Single Oral Dose of Ritonavir on the Single Dose Pharmacokinetics of ASP2151 in Healthy Men
Brief Title: Drug-Drug Interaction Study: ASP2151 and Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: M522101-EU22; 2014-002174-37 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-22 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: HSV; HIV; Herpes; volunteers; drug-drug interaction
MeSH Terms: conditions — Herpes Simplex | interventions — ASP2151; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400mg ASP2151 (Other): 400mg ASP2151 alone followed by 400mg ASP2151 + 600mg ritonavir
  Interventions: Drug: ASP2151; Drug: ritonavir
- 1200mg ASP2151 (Other): 1200mg ASP2151 alone followed by 1200mg ASP2151 + 600mg ritonavir
  Interventions: Drug: ASP2151; Drug: ritonavir

INTERVENTIONS:
Drug: ASP2151
Drug: ritonavir
  Other Names: Norvir

SUMMARY:
ASP2151 is an experimental treatment for herpes. HIV infected people are susceptible to contracting other infections because of their compromised immune system. As HIV patients will be taking drugs to treat the virus this study aims to see if ASP2151 would interact with one of the drugs that is commonly prescribed to HIV patients (ritonavir).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Any of the following liver function tests higher than 1.5 times the ULN at the screening visit: aspartate aminotransferase (AST), alanine aminotransferase (ALT), ALP, bilirubin, gamma glutamyl transpeptidase (gamma-GT).
* Platelet counts outside normal limits.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Clinically significant impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* History of bleeding diathesis.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of severe adverse reaction to any drug, history of multiple drug allergies (multiple defined as >3), or sensitivity to trial medication.
* Use, during the 28 days before the first dose of trial medication, of any prescription medicine, or any other medicine or herbal remedy (such as St John's wort) known to interfere with the CYP3A4 metabolic pathway (unless judged as not clinical significant by the investigator and sponsor).
* Use, during the 7 days before the first dose of trial medication, of any over-the-counter medicine, with the exception of paracetamol (acetaminophen).
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 10 cigarettes daily.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Blood pressure (BP) and heart rate (HR) in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40_100 beats/min.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in United Kingdom from 05-September 2014 to 04-December 2014
Groups:
- 400mg ASP2151: ASP2151 400mg alone followed by ASP2151 400mg + 600 mg ritonavir, or vice versa.
- 1200mg ASP2151: ASP2151 1200mg alone followed by ASP2151 1200mg + 600 mg ritonavir, or vice versa.
Period: Overall Study
Arm/Group | 400mg ASP2151 | 1200mg ASP2151
Started | 24 | 24
First Intervention (8 Days) | 24 | 24
Wasout (2weeks) | 24 | 24
Second Intervention (8 Days) | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400mg ASP2151 | 1200mg ASP2151 | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 28.2 (6.4) | 27 (4.9) | 27.6 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 24 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 21 | 24 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 17 | 15 | 32
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of ASP2151
Time Frame: Blood samples were taken at pre-dose of Day 1 and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72h after post doses in first or second intervention
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 400 mg ASP2151 Alone: ASP2151(400 mg) alone
- 400mg ASP2151 With Ritonavir: 400mg ASP2151 alone followed by 400mg ASP2151 + 600mg ritonavir
  ASP2151
  ritonavir
- 1200 mg ASP2151 Alone: ASP2151(1200 mg) alone
- 1200mg ASP2151 With Ritonavir: 1200mg ASP2151 alone followed by 1200mg ASP2151 + 600mg ritonavir
  ASP2151
  ritonavir
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 1845.7 (25.4) | 2518.7 (21.9) | 3804 (28.8) | 6211.6 (29.2)

2. Primary Outcome: Time of Peak Concentration (Tmax) of ASP2151
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 3 [1.00 to 4.00] | 4 [1.00 to 10.00] | 3.025 [1.00 to 4.12] | 4 [2.00 to 12.00]

3. Primary Outcome: Area Under the Curve (AUC) of ASP2151
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 23162.4 (34.2) | 60225.3 (23) | 48532.3 (29.3) | 162131.6 (25.3)

4. Primary Outcome: Half-Life (t1/2) of ASP2151
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 7.375 (14.9) | 12.575 (15.9) | 7.178 (17.5) | 12.498 (19.6)

5. Primary Outcome: Apparent Total Body Clearance (CL/F) of ASP2151 From Plasma
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
L/h | 18.314 (7.2654) | 6.815 (1.6607) | 25.735 (7.5753) | 7.63 (1.9843)

6. Primary Outcome: Apparent Volume of Distribution (Vd/F) of ASP2151
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
L | 190.1 (56.912) | 123.17 (28.366) | 266.33 (79.948) | 139.33 (43.231)

7. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Refer to the result of adverse event.
Time Frame: Up to 31 days
Measure: Number; unit: participants
Groups:
- 400 mg ASP2151 Alone: 400 mg ASP2151 alone
- 400 mg ASP2151 With Ritonavir: 400 mg ASP2151 with 600 mg ritonavir
- 1200 mg ASP2151 Alone: 1200 mg ASP2151 alone
- 1200 mg ASP2151 Withritonavir: 1200 mg ASP2151 with 600 mg ritonavir
Arm/Group | 400 mg ASP2151 Alone | 400 mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200 mg ASP2151 Withritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants
  Non-serious adverse event | 8 | 17 | 15 | 13
  serious adverse event | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 189.9 (27.7) | 21.6 (70.7) | 421.5 (36.7) | 56.2 (79.9)

9. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 3 [1.00 to 4.07] | 1.5 [1.00 to 12.07] | 3 [1.98 to 6.00] | 1.01 [0.5 to 23.98]

10. Other Pre Specified Outcome: Area Under the Curve (AUC) of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 2636.2 (25.8) | 744.4 (12) | 6023.1 (30.2) | 1646.1 (37.3)

11. Other Pre Specified Outcome: Half-life (t1/2) of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 8.063 (18.1) | 40.213 (56.6) | 7.617 (18.6) | 42.197 (69.1)

12. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/F) From Plasma of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
L/h | 156.72 (43.197) | 540.93 (68.554) | 207.45 (59.311) | 775.35 (315.166)

13. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/F) of ASP1955888-00
Description: ASP1955888-00 is a metabolite of the study drug (ASP2151)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 400 mg ASP2151 Alone | 400mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200mg ASP2151 With Ritonavir
Number analyzed (Participants) | 24 | 24 | 24 | 24
L | 1840.8 (559.49) | 21474 (4135.72) | 2340.7 (877.14) | 27624.2 (14413.73)

ADVERSE EVENTS:
Time Frame: Up to 31 days after the final dose
Groups:
- 1200 mg ASP2151 With Ritonavir: 1200 mg ASP2151 with 600 mg ritonavir
Arm/Group | 400 mg ASP2151 Alone | 400 mg ASP2151 With Ritonavir | 1200 mg ASP2151 Alone | 1200 mg ASP2151 With Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 8/24 | 17/24 | 15/24 | 13/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 mg ASP2151 Alone (N=24) | 400 mg ASP2151 With Ritonavir (N=24) | 1200 mg ASP2151 Alone (N=24) | 1200 mg ASP2151 With Ritonavir (N=24)
Headache (Nervous system disorders) | 3 | 6 | 8 | 7
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No